CLINICAL TRIAL: NCT04307277
Title: Interest of Peri Operative CHemotherapy In Patients With CINSARC High-risk Localized Soft Tissue Sarcoma
Acronym: CHIC-STS01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19SARC05
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma; CINSARC signature; Chemotherapy
MeSH Terms: conditions — Sarcoma | interventions — Standard of Care; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Other)
  Interventions: Other: Standard of care
- Experimental arm (Experimental)
  Interventions: Drug: Standard of care + chemotherapy

INTERVENTIONS:
Drug: Standard of care + chemotherapy — Doxorubicine with Ifosfamide during 4 cycles Q3W Or Doxorubicine with Dacarbazine during 4 cycles Q3W (for patients with Leiomyosarcoma)
  Arms: Experimental arm
Other: Standard of care — Surgical excision with external radiotherapy (if applicable)
  Arms: Control arm

SUMMARY:
Phase III, multicenter, randomized open-label and comparative study designed to demonstrate whether adding 4 cycles of peri-operative doxorubicin-based chemotherapy improves metastasis-free survival as compared with standard management in patients with resectable STS, considered as high-risk according to CINSARC (Complexity Index in SARComas) signature.

After signed informed consent, patients considered as eligible to CHIC-STS study by the investigator will be enrolled in the study and a molecular screening will be performed (600 patients will be screened).

Patients considered as low-risk according to CINSARC signature will be treated at the discretion of the clinicians (prospective cohort).

Patients considered as high-risk according to CINSARC signature will be randomized in the open-label multicenter phase III trial and assigned in one of the two following treatments arms:

* Arm A (control arm): Standard of care (surgical excision +/- external radiotherapy).
* Arm B (experimental arm): Standard of care + 4 cycles of intravenous chemotherapy during 12 weeks.

A total of 250 patients will have to be randomized with 125 patients in each arm.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of soft-tissue sarcoma, histologically confirmed by RRePS (Réseau de Référence en Pathologie des Sarcomes et des Viscères) network
2. According to FNCLCC grading system, grade 1, 2 or 3 tumors
3. Resectable and localized disease after appropriate extension work-up (including at least a chest-CT)
4. 6 weeks or less between surgical excision and inclusion (if performed before inclusion)
5. Available archived FFPE tumor sample in sufficient quantity to allow CINSARC qualification
6. Age ≥ 18 years
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
8. Life expectancy of at least 12 weeks after the start of the treatment
9. Women should be post-menopaused or willing to accept the use of an effective contraceptive regimen during the treatment period and at least 12 months (ifosfamide treatment) or 6 months (dacarbazine treatment) after the end of the treatment period. All non-menopaused women should have a negative pregnancy test within 72 hours prior to registration. Men should accept to use an effective contraception during treatment period and at least 3 months after the end of the study treatment.
10. Signed written informed consent
11. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Soft-tissue sarcoma with the following histological subtypes: well-differentiated liposarcomas, alveolar soft-part sarcoma, dermatofibrosarcoma protuberans, clear-cell sarcoma, epithelioid sarcoma, alveolar or embryonal rhabdomyosarcoma
2. Primitive cutaneous, retroperitoneal, uterus or visceral STS
3. Metastatic disease
4. Previous or ongoing treatment for the sarcoma (with the exception of surgical excision)
5. Contra-indication for Doxorubicin, Ifosfamide and Dacarbazine treatments
6. Prior therapy with ifosfamide or cyclophosphamide or other nitrogen mustards, and prior therapy with anthracyclines
7. Prior mediastinal/cardiac radiotherapy
8. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia, myocardial infarction within 6 months prior to study entry
9. Prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma
10. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
11. Known infection with HIV, hepatitis B, or hepatitis C
12. Women who are breastfeeding, pregnant or who plan to become pregnant while in the trial
13. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
14. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice)
15. Patient unable to comply with the protocol for any reason.

ADDITIONAL CRITERIA FOR THE RANDOMIZED PHASE III STUDY

1. High-risk CINSARC signature
2. Acceptable hematologic function (within 72 hours prior randomization): Absolute neutrophil count (ANC) ≥ 1.5 G/L, Platelet count ≥ 100 G/L and Hemoglobin > 9g/dL
3. Acceptable renal function within 72 hours prior randomization: Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 60 mL/min (by the Cockcroft and Gault formula)
4. Acceptable liver function: Bilirubin ≤ 1.5 x upper limit of normal (ULN), AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN
5. Normal LVEF (>50%) measured by echocardiography or isotopic ventriculography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2032-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival defined by the delay between randomization and the appearance of metastatic. | 5 years for each patient

SECONDARY OUTCOMES:
Disease-free survival defined by the delay between randomization and first relapse (local, regional, or distant) or death from any cause. | 5 years for each patient
Safety assessed by the toxicity grading of the National Cancer Institute (NCI-CTCAE v5.0). | 4 months for each patient
Overall survival defined by the delay between randomization and death from any cause. | 5 years for each patient

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - CHRU Besançon, Besançon
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-François Leclerc, Dijon
  - CHU Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHU Marseille, Marseille
  - Institut de Cancérologie de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hôpital Cochin, Paris
  - CHU Poitiers, Poitiers
  - Institut Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - Institut de Cancérologie de Lorraine - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Filleron T, Le Guellec S, Chevreau C, Cabarrou B, Lesluyes T, Lodin S, Massoubre A, Mounier M, Poublanc M, Chibon F, Valentin T. Value of peri-operative chemotherapy in patients with CINSARC high-risk localized grade 1 or 2 soft tissue sarcoma: study protocol of the target selection phase III CHIC-STS trial. BMC Cancer. 2020 Jul 31;20(1):716. doi: 10.1186/s12885-020-07207-3. PMID 32736540